CLINICAL TRIAL: NCT01500707
Title: A Single Dose Study to Assess the Pharmacokinetics of SCH 900800 Administered as Oral Tablets in L-DOPA-treated Subjects With Parkinson's Disease
Brief Title: Single Dose Study to Assess the Pharmacokinetics of SCH 900800 in Subjects With Parkinson's Disease Being Treated With Levodopa (L-DOPA) (P08235)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P08235
Record Dates: First submitted 2011-12-22; First posted 2011-12-28 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SCH 900800 (Experimental): Participants receiving a single dose of SCH 900800
  Interventions: Drug: SCH 900800

INTERVENTIONS:
Drug: SCH 900800 — SCH 900800, one 20 mg tablet, orally
  Other Names: MK-8800

SUMMARY:
This study is being done to assess the pharmacokinetics of SCH 900800 in participants with moderate to severe Parkinson's Disease (PD) being treated with L-DOPA.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 18 and 35
* Diagnosis of idiopathic Parkinson's disease (PD) characterized by at least two of the following: resting tremor, bradykinesia, rigidity (must have either resting tremor or bradykinesia); participants must have either moderate severity PD or moderate to severe PD with motor fluctuations
* For participants with moderate PD, Hoehn and Yahr stage must be ≥1.5 and ≤4 in the "off" state at Screening; for participants with moderate to severe PD with motor fluctuations, Hoehn and Yahr stage must be ≥2 and ≤4 in the "on" state at Screening
* On stable anti-parkinson treatment regimen that includes L-DOPA/carbidopa for at least 3 weeks prior to screening and clinically stable at the time of randomization (predose), and first morning dose of L-DOPA must be 100 mg or greater
* L-DOPA therapy for ≥ 6 months prior to screening
* If taking adjunct PD medications (amantadine, anticholinergics, DOPA decarboxylase inhibitor, dopamine agonist, entacapone, rasagiline or selegiline) must be on stable dose for at least 4 weeks prior to randomization on this study
* Females, if fertile, willing to use a medically acceptable method of contraception for 3 months prior to screening through 2 months after stopping study drug
* Non-vasectomized males must agree to use a condom with spermicide (when

marketed in the country) or abstain from sexual intercourse during the trial and for 3 months after stopping the study drug

Exclusion Criteria:

* Pregnant or intending to become pregnant within 3 months of ending study therapy
* Breastfeeding
* Systolic blood pressure (BP) ≥150 mm Hg or diastolic BP ≥90 mm Hg at Screening and at a BP recheck prior to randomization. If antihypertensive medications are used to control BP, dose of antihypertensive medications must be stable for at least 2 weeks prior to randomization
* History of clinically significant cardiovascular disease or procedure prior to randomization, including, but not limited to, myocardial infarction, prolonged QT interval corrected for heart rate, other clinically important ECG abnormality, angioplasty, stable or unstable angina, or heart failure
* History of clinically significant or uncontrolled neurologic (other then Parkinson's disease) endocrine, gastrointestinal, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases
* Surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of any drug including history or presence of inflammatory bowel disease, ulcers, gastrointestinal or rectal bleeding; history of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection; history of pancreatic injury or pancreatitis; history or presence of liver disease or liver injury; history or presence of impaired renal function as indicated by clinically significant elevation in creatinine, blood urea nitrogen (BUN)/urea, urinary albumin, or clinically significant urinary cellular constituents ; or history of urinary obstruction or difficulty in voiding
* Infectious disease within 4 weeks prior to drug administration
* Positive for hepatitis B surface antigen, hepatitis C antibodies or human immunodeficiency virus (HIV)
* Clinically significant complications of Parkinson's disease or Parkinson's disease treatments, including severe, disabling motor fluctuations that do not allow the subject to maintain a stable L-DOPA/carbidopa dose; disabling dyskinesias; hallucinations; or dementia
* History of alcohol or drug abuse in the past 2 years
* Donation of blood in the past 60 days
* Previously received SCH 900800
* Currently participating in another clinical study or participated in a clinical study in which an investigational drug or surgical procedure was administered, within 30 days of baseline
* Study staff personnel or family members of the study staff personnel
* Use of more than 10 cigarettes or equivalent tobacco use per day
* History of malignancy
* A form of parkinsonism other than idiopathic Parkinson's disease (e.g., multiple system atrophy or progressive supranuclear palsy)
* Imminent risk of self-harm or of harm to others, based on clinical interview and responses on the Columbia Suicidality Severity Rating Scale. Exclude any participant reporting suicidal ideation with intent, with or without a plan in the past 2 months or suicidal behavior in the past 6 months
* Use of strong or moderate inhibitors or inducers of cytochrome P (CYP) 3A4 isoenzyme (e.g. St John's Wort, ketoconazole, ritonavir, rifampin, macrolide antibiotics, some calcium channel blockers including diltiazem, verapamil, etc.) within 30 days; inhibitors of enzyme CY2D6 within 14 days; Proton Pump Inhibitors or histamine (H2) Receptor Blockers within 14 days

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Area under the concentration time curve from Hour 0 to infinity (AUC0-∞) of SCH 900800 | Hour 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 14, 32, 48, 72, and 96 hours post-dose
Maximum concentration (Cmax) of SCH 900800 | Hour 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 14, 32, 48, 72, and 96 hours post-dose